CLINICAL TRIAL: NCT05362357
Title: iSTART: A Campus & Community Initiative for Services in Tec-health
Acronym: iSTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Northridge (Other)
Responsible Party: Principal Investigator, Bethany Rainisch, Principal Investigator, Associate Professor, California State University, Northridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H79SP021733
Record Dates: First submitted 2022-04-28; First posted 2022-05-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Substance Use; Binge Drinking; Marijuana Use; Alcohol Drinking; Prescription Opioid Misuse; Illicit Drug Use
Keywords: Web-app; Module; mHealth
MeSH Terms: conditions — Substance-Related Disorders; Binge Drinking; Marijuana Use; Alcohol Drinking; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prevention Group (Experimental): Web-app with five weekly substance modules. Each module is approximately 15 minutes long.
  Interventions: Behavioral: iSTART Web-app
- Comparison Group (Active Comparator): Web-app with single abbreviated module combining all five substances. Module is approximately 20 minutes long.
  Interventions: Behavioral: iSTART Web-app
- Control Group (No Intervention): No access to web-app.

INTERVENTIONS:
Behavioral: iSTART Web-app — 30-day substance prevention web-app for students at a Hispanic Serving Institution.
  Arms: Comparison Group; Prevention Group

SUMMARY:
The iSTART intervention is a 30-day substance prevention web-app whereby students complete five weekly interactive modules using a smart device or computer. Each module is approximately 15 minutes long, and focuses on a select substance: (i) alcohol, (ii) marijuana, (iii) nicotine, (iv) prescription drugs, and (v) illicit drugs. The modules are based on key theoretical constructs, behavior change strategies, and practical module components: attitudes (knowledge), perceived susceptibility (risk perceptions), subjective norms (normative re-education), and self-efficacy (refusal skills). This intervention will be evaluated via a time series design using a sample of 600 students randomly assigned to either the intervention, comparison, or control condition at a public institution in southern California.

ELIGIBILITY:
Inclusion Criteria:

* Current Cal State Northridge (CSUN) matriculated students
* Age 18-30

Exclusion Criteria:

* Not currently a CSUN student
* Not 18-30 years of age
* Identified as having an alcohol or substance use disorder (AUD or SUD) as determined by the brief DSM-5 screener

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1100 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline alcohol use behavior at 3 months. | Baseline and 90-days following intervention completion.
  Measured as the number of days drinking alcohol in past 30-days
Change from baseline binge drinking at 3 months. | Baseline and 90-days following intervention completion.
  Measured as the number of days consumed five or more alcoholic beverages at the same time for males; four or more for females in past 30-days.
Change from baseline tobacco use at 3 months. | Baseline and 90-days following intervention completion.
  Measured as the number of days using cigarettes, pipe tobacco, chewing tobacco, snus in past 30-days.
Change from baseline electronic vaping at 3 months. | Baseline and 90-days following intervention completion.
  Measured as the number of days vaped in past 30-days.
Change from baseline marijuana use at 3 months. | Baseline and 90-days following intervention completion.
  Measured as the number of days smoked marijuana in past 30-days.
Change from baseline non-prescribed prescription drug use at 3 months. | Baseline and 90-days following intervention completion.
  Measured as the number of days used stimulants, sedatives, benzodiazepines, and prescription opioids in past 30-days.
Change from baseline illicit drug use at 3 months. | Baseline and 90-days following intervention completion.
  Measured as the number of days used cocaine, amphetamines, MDMA/Ecstasy, heroin, fentanyl, and non-Rx opioids in past 30-days.

SECONDARY OUTCOMES:
Change from baseline behavioral intent at 3 months. | Baseline and 90-days following intervention completion.
  Measured as the intent to smoke marijuana/cigarettes, binge drink, and use non-prescribed drugs. Participants are asked to rate the likelihood of use in the next 30 days on a four-point Likert scale from 1=very likely to 4=very unlikely.
Change from baseline alcohol-specific outcomes at 3 months. | Baseline and 90-days following intervention completion.
  Measured as participants who report any past 30-day alcohol use indicate how many times they have experienced ten select outcomes in the last 30 days while drinking alcohol, or as the result of their alcohol use. Example items include: 'Not being able to do your homework or study for a test', 'Missed out on other things because you spent too much money on alcohol', 'Went to work or school high or drunk', 'Felt that you needed more alcohol than you used to use in order to get the same effect', and 'Had withdrawal symptoms, that is, felt sick because you stopped or cut down on drinking'. Participants respond: 'never', '1-2 times', '3-5 times', '6-10 times', and 'more than 10 times' in the past 30-days.

OTHER OUTCOMES:
Change from baseline risk perceptions at 3 months. | Baseline and 90-days following intervention completion.
  Measured by participants' evaluation of their perceived risk level for the following six substance use behaviors: binge drinking once or twice a week, tobacco use once or twice a week, marijuana use once or twice a week, prescription opioid use once or twice a week, non-prescription opioid use once or twice a week, sharing needles/injection equipment, injecting drugs, and illicit drug use. Response options for each behavior include 1='no risk', 2='slight risk', 3='moderate risk', 4='great risk', or 9='don't know'.
Change from baseline subjective norms at 3 months. | Baseline and 90-days following intervention completion.
  Measured by participants' indication of what percentage of students on campus they perceive use a variety of substances within the last 30 days, (i.e., alcohol, cigarettes, marijuana, different prescription drugs, and several illicit drugs) choosing one of ten percentile intervals from 0-100%.
Change from baseline refusal self-efficacy at 3 months. | Baseline and 90-days following intervention completion.
  Self-efficacy will be evaluated through two refusal skills statements: "I would be able to say no if a friend offered me a drink of alcohol" and "I would be able to refuse if a friend offered me drugs, including marijuana", by indicating their level of agreement on a four-point Likert scale from 1='strongly agree' to 4='strongly disagree'.
Socio-demographics | Baseline
  Participant characteristics, including age, Hispanic origin, race, sex at birth, gender identification, sexual orientation, living situation, college status, military service/veteran status, arrest history, parole/probation status, and household income
Adverse Childhood Experiences (ACE) | Baseline
  ACE are conceptualized as maltreatment (e.g., verbal, emotional, physical, and sexual abuse), and household dysfunction (e.g., parent/caregiver substance use, intimate partner violence, incarceration, homelessness, mental illness, separation/divorce (71). Participants respond to each of the ten ACE items as 1=Yes or 0=No. An ACE score will be computed with a range from 0-10.
Developmental transition | Baseline
  Participants respond 1=Yes or 0=No to a list of 18 major life events within the last three years. Example life events include: getting into a new romantic relationship; breaking up with a girlfriend or boyfriend; losing a job; being unemployed and not able to find work; caring for a parent or relative; getting extremely ill; having a baby; losing a baby; or having family separated due to immigration. A total score will be computed with a range from 0-18.

CONTACTS AND LOCATIONS:
Locations (1):
- California State University, Northridge, Northridge, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once the study is complete, the PI and evaluator will determine whether IPD will be made available to other researchers beyond traditional research dissemination via peer-reviewed journal articles and conference presentations.

REFERENCES:
- [Derived] Rainisch BKW, Dahlman L, Vigil J, Forster M. Using a multi-module web-app to prevent substance use among students at a Hispanic Serving Institution: development and evaluation design. BMC Public Health. 2022 Jun 15;22(1):1198. doi: 10.1186/s12889-022-13428-x. PMID 35705975